CLINICAL TRIAL: NCT01043003
Title: Support for Hispanic Breast Cancer Patients and Caregivers
Brief Title: Bilingual Breast Cancer Educational Intervention for Hispanic Women With Stage I, Stage II, or Stage III Breast Cancer and Their Families or Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 06136; NCI-2009-01548
Record Dates: First submitted 2010-01-04; First posted 2010-01-06 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-06

CONDITIONS: Breast Cancer; Ductal Breast Carcinoma in Situ; Stage I Breast Cancer; Stage II Breast Cancer; Stage IIIA Breast Cancer; Stage IIIB Breast Cancer; Stage IIIC Breast Cancer
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Intraductal, Noninfiltrating | interventions — Early Intervention, Educational; Methods; Psychiatric Rehabilitation; Caregivers

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (Experimental): Patients and caregivers undergo the Bilingual Breast Cancer Educational Intervention (BBCEI) comprising teaching sessions over 50-65 minutes about 4 specific domains (i.e., physical, psychological, social, and spiritual well being) once weekly during month 1 and also undergo evaluation sessions at months 1, 4, and 7. Patients and caregivers receive reinforcement telephone calls every other week.
  Interventions: Other: educational intervention; Procedure: quality-of-life assessment; Other: Questionnaire Administration; Other: psychosocial support for caregiver; Procedure: assessment of therapy complications; Other: informational intervention
- Arm II (Active Comparator): Patients and caregivers undergo usual care comprising evaluation sessions at months 1, 4, and 7. Patients and caregivers may undergo the 4 BBCEI teaching sessions during month 7. Patients and caregivers receive reinforcement telephone calls every other week.
  Interventions: Procedure: quality-of-life assessment; Other: Questionnaire Administration; Other: psychosocial support for caregiver; Procedure: assessment of therapy complications; Other: informational intervention

INTERVENTIONS:
Other: educational intervention — Undergo Bilingual Breast Cancer Educational Intervention
  Other Names: intervention, educational
  Arms: Arm I
Procedure: quality-of-life assessment — Ancillary studies
  Other Names: quality of life assessment
Other: Questionnaire Administration — Ancillary studies
Other: psychosocial support for caregiver — Support for caregiver
Procedure: assessment of therapy complications — Ancillary study
Other: informational intervention — Undergo evaluation sessions

SUMMARY:
RATIONALE: Studying quality-of-life in patients having cancer treatment may identify the intermediate- and long-term effects of treatment on patients with cancer

PURPOSE: This randomized clinical trial is studying how well an educational intervention works in supporting Hispanic women with stage I, stage II, or stage III breast cancer and their families or caregivers.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Test the effects of the Bilingual Breast Cancer Education Intervention (BBCEI) on outcomes of breast cancer survivors (BCS) and family caregivers at 1, 3, and 6 months post intervention.

II. Test the effect of influencing demographic and treatment variables on outcomes of the BBCEI at 1, 3, and 6 months post intervention.

III. Examine the perceived quality of the BBCEI.

OUTLINE: Patients and caregivers are randomized to 1 of 2 intervention arms.

ARM I: Patients and caregivers undergo the Bilingual Breast Cancer Educational Intervention (BBCEI) comprising teaching sessions over 50-65 minutes about 4 specific domains (i.e., physical, psychological, social, and spiritual well being) once weekly during month 1 and also undergo evaluation sessions at months 1, 4, and 7.

ARM II: Patients and caregivers undergo usual care comprising evaluation sessions at months 1, 4, and 7. Patients and caregivers may undergo the 4 BBCEI teaching sessions during month 7.

All patients and caregivers receive reinforcement telephone calls every other week.

ELIGIBILITY:
Inclusion

* Histologically confirmed diagnosis of stage 0 (DCIS), I, II, or III breast cancer
* No evidence of recurrent, metastatic, or second primary cancer
* Completing primary treatment with surgery, radiation therapy (if indicated), and/or adjuvant chemotherapy (if indicated)
* Subjects may be on hormonal therapy after treatment for initial breast cancer
* Self-identification as Hispanic/Latino
* Able to read and understand English or Spanish to participate in the patient teaching
* Able and willing to participate in the study
* The Caregiver selection criteria is: self-identification as the primary caregiver; age 18 years or over; self-identification as Hispanic/Latino; Able to read and speak English or Spanish; Able and willing to participate in the study

Exclusion

* Patients will be excluded if they are actively receiving treatment with surgery, radiation therapy, or chemotherapy; patients may be receiving adjuvant hormonal therapy such as Tamoxifen during the course of the study since it is recommended for five years after primary and adjuvant therapy
* Patients who have recurrence, metastasis, or a second primary cancer will not be recruited for the study; if however, they develop recurrence, metastasis, or a second primary cancer during the time of the study participation, the subjects will remain in the study
* Patients will not be recruited directly from support groups because of potential bias inherent in sample attending support groups; however, some patients may be participating in support groups or other forms of counseling

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2006-08; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Effects of the Bilingual Breast Cancer Education Intervention on outcomes (physical, psychological, social, spiritual, and overall quality of life) of breast cancer survivor and family caregivers | At 1, 3, and 6 months post intervention
Effect of influencing demographic and treatment variables on outcomes of the BBCEI | At 1, 3, and 6 months post intervention
Perceived quality of the BBCEI | At 1, 3, and 6 months post intervention

CONTACTS AND LOCATIONS:
Overall Officials: Gloria Juarez, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope, Duarte, California, United States